CLINICAL TRIAL: NCT00357864
Title: Basic Research on Carbachol´s Headache Inducing Characteristics and Effects on the Cerebral Blood Flow in a Humane Experimental Headache Model
Brief Title: Carbachol´s Headache Inducing Characteristics and Effects on the Cerebral Blood Flow
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Other Study IDs: 2006-002462-19
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2007-08

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Carbachol

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carbachol

SUMMARY:
To investigate headache score and accompanying symptoms during and after infusion of carbachol.

DETAILED DESCRIPTION:
To investigate headache score and accompanying symptoms during and after infusion of carbachol.

Changes in regional cerebral blood flow (rCBF) in the area supplied by middle cerebral artery (MCA), blood flow in MCA, diameter of the superficial temporal artery (STA) and radial artery (RA)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-40
* 50-100 kg
* Fertile women must use safe contraceptives (IUD, oral contraceptives, surgical sterilisation and long lasting gestagen.

Exclusion Criteria:

* Tension type headache more than once/month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the halflife for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Headache within the last 24 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-07; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: henrik schytz, Principal Investigator — Danish Headache Center
Locations (1):
- Dansih Headache Center, Glostrup Municipality, Denmark